CLINICAL TRIAL: NCT02299947
Title: Comparison of a Single Dose Fibrinogen With Placebo and the Number of Blood Transfusions After Ascending Aorta Surgery (FIBTEG Study)
Brief Title: Bloodtranfusions After Aortic Surgery
Acronym: FIBTEG
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow inclusion
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, dr. P. Noordzij, MD PhD, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL45370.100.14
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Hemorrhage; Thoracic Aneurysm
MeSH Terms: conditions — Hemorrhage; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Haemocomplettan P (Experimental): Study patients that receive Haemocomplettan P
  Interventions: Drug: Haemocomplettan P
- NaCl 0.9% (Placebo Comparator): Study patients that receive NaCl 0.9%
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Haemocomplettan P
  Arms: Haemocomplettan P
Drug: Placebo
  Arms: NaCl 0.9%

SUMMARY:
The purpose of this study is to answer the following question: Leads a primary coagulation corrected with a single dose of fibrinogen concentrate after ascending aorta-arc reconstruction to a decrease in the number of allogenic blood transfusions, compared to placebo?

DETAILED DESCRIPTION:
Cardiothoracic surgery (CTC) is associated with blood loss and an increased risk for impaired coagulation by the use of a CBP. Coagulation is a process of primary hemostasis by adhesion of trombocytes and aggregation, followed by secondary coagulation and fibrin formation. During CTC fibrinogen is the first coagulation factor which reaches critical concentration necessary for clotting. Point of Care clotting assay with thromboelastography (TEG) provides qualitative information on coagulation factors and clot strength. Specific coagulation factor correction of impaired clotting improves clot strength and may reduces the number of perioperative allogeneic blood transfusions, resulting in possible reduction of postoperative blood loss and reduction of the risk of re-operation in the short and long term. The hypothesis of this study is that a single dose fibrinogen concentrate immediately after CTC leads to a decrease in the number of allogenic blood transfusions in patients with clinically impaired clotting, verified by TEG.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery for thoracic aneurysm

Exclusion Criteria:

* Prior trombosis or myocardial infarction, congenital coagulation disorder, use of anti-coagulants prior to surgery, prior thoracic surgery, pregnancy, pre-operative fibrinogen concentration <1g/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
Number of transfused blood products | 24 hours after surgery

SECONDARY OUTCOMES:
Blood loss | 24 hours after surgery
Re-operation | 30 day after surgery
Mortality | 30 day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Peter Noordzij, PhD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St Antonius hospital, Nieuwegein, Utrecht, Netherlands